CLINICAL TRIAL: NCT00195520
Title: An Open Assessment of the Effect of Low-Dose Totelle® 1 mg on Menopausal Symptoms, Sexual Function and Quality of Life
Brief Title: Study Evaluating Totelle® in Menopausal Symptoms and Sexual Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0753T-101537
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Hot Flashes; Sleep Disorders
Keywords: Menopause; Sleep Disorder; Hot Flashes
MeSH Terms: conditions — Hot Flashes; Sleep Wake Disorders

INTERVENTIONS:
Drug: Totelle®

SUMMARY:
To evaluate the tolerability, bleeding patterns and acceptability of Totelle® 1mg administered to a population of Brazilian women in a continuous combined regime for hormone replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Intact uterus
* Generally health postmenopausal women 45 to 60 years of age, inclusive
* Sexually active
* No hormone replacement therapy within the 90 days immediately prior to the screening evaluation.

Exclusion Criteria:

* Known or suspect estrogen-dependent neoplasia
* Known hypersensitivity to estrogens, progestins, or other ingredients of Totelle
* Use of any estrogen, progestin, androgen containing medications or tibolone within 12 weeks before screening.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-12; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the tolerability, bleedeing patterns and acceptability of Totelle 1mg administered to a population of Brazilian women in a continuous combined regime for hormone replacement therapy.

SECONDARY OUTCOMES:
To evaluate the effects of Totelle 1 mg on sexual function and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (2):
- Brazil (2):
  - Jundiaí, São Paulo
  - São Paulo, São Paulo